CLINICAL TRIAL: NCT04349215
Title: Validation of the Chinese Version of the Obstetric Quality of Recovery Scoring Tool (ObsQoR-11) at Early and Intermediate Phases After Elective Caesarean Delivery: a Multicentre Observational Trial
Brief Title: Validation of the Chinese ObsQoR-11
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002016RINC
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2020-04

CONDITIONS: Cesarean Delivery
Keywords: Cesarean delivery,the Obstetric Quality of Recovery-11 score, Chinese

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigation of post-cesarean recovery among Taiwanese pregnant women.

DETAILED DESCRIPTION:
Improving postpartum quality of recovery is important particularly for women undergoing cesarean delivery. This is because cesarean delivery is associated with significant postoperative pain and risks of anesthesia-related adverse effects. To improve the quality of recovery after a cesarean delivery, the first step is to find out the most relevant perioperative factors.

In response to this problem, experts including anesthesiologists, obstetricians and midwives from University College London Hospital, Royal Free Hospital, London as well as Stanford University established a set of 11-item questionaire related to postpartum recovery, namely the Obstetric Quality of Recovery-11 score (ObsQoR-11), with a total score of 110. The latest systemic review in 2020 also confirmed that this questionnaire is the best option for recovery assessment after cesarean delivery. However, for women undergoing cesarean delivery in Taiwan, it is still unknown whether this questionnaire is representative or not. Therefore, this study aims to include women undergoing elective cesarean delivery from three hospitals in Taiwan.

ELIGIBILITY:
Inclusion criteria

1. age>= 20 yr
2. elective cesarean delivery

Exclusion:

emergent surgery

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Post-cesarean delivery recovery
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Validation of the Chinese ObsQoR-11 score | 5 days
  To validate the Chinese ObsQoR-11 at 24 hour and 96 hour after cesarean delivery

SECONDARY OUTCOMES:
Assessment of reliability, acceptability, and responsiveness of the Chinese ObsQoR-11 | 5 days
  Perform analysis of reliability, acceptability, and responsiveness test for the Chinese ObsQoR-11

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital; Cathay General Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan